CLINICAL TRIAL: NCT01486498
Title: Health Economic Analyses of Treatment Strategies for Allergic Respiratory Diseases
Brief Title: Quality of Life and Health Economic Measurements in Allergic Patients Treated With Immunotherapy
Acronym: SABAL
Status: Completed | Type: Observational
Sponsor: Aalborg University (Other)
Responsible Party: Principal Investigator, Karin Dam Petersen, Associate Professor, Aalborg University
Other Study IDs: SABAL
Record Dates: First submitted 2011-12-03; First posted 2011-12-06 (Estimated); Last update posted 2011-12-06 (Estimated); Status verified 2011-12

CONDITIONS: Hypersensitivity; Asthma; Rhino-Conjunctivitis; Quality of Life; Effects of Immunotherapy
MeSH Terms: conditions — Hypersensitivity; Asthma

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Grass pollen and house dust mites (HDM) are the most common allergens causing allergic rhino-conjunctivitis (RC) and/or asthma (A). Subcutaneous allergen specific immunotherapy (SCIT) reduces symptoms and use of medication. The purpose of SABAL is to assess the effect of SCIT on disease severity classifications in terms of number of days affected- and sick days on patients with grass pollen and/or HDM induced disease. These outcome measures will be gathered in one single measure: Quality Adjusted Life Years (QALY)

ELIGIBILITY:
Inclusion Criteria:

* Adults (> 16 years) and allergic to grass pollen and/or house dust mites.

Exclusion Criteria:

* Allergic patients who had been immunotherapy treated before.

Min Age: 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: The intervention group consisted of 254 patients receiving subcutaneous allergen specific immunotherapy (SCIT) with grass pollen and/or house dust mite extracts. The control group consisted of 317 patients with grass pollen and/or house dust mite allergy, who were not receiving SCIT.
Sampling Method: Non-Probability Sample
Enrollment: 571 (Actual)
Dates: Start 2005-11; Primary Completion 2009-11 (Actual); Study Completion 2011-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Karin D Petersen, PhD, Study Chair — Associate Professor

REFERENCES:
- [Derived] Petersen KD, Kronborg C, Larsen JN, Dahl R, Gyrd-Hansen D. Patient related outcomes in a real life prospective follow up study: Allergen immunotherapy increase quality of life and reduce sick days. World Allergy Organ J. 2013 Sep 9;6(1):15. doi: 10.1186/1939-4551-6-15. PMID 24229439